CLINICAL TRIAL: NCT01537055
Title: Comparison of the Efficacy of Levofloxacin-based Sequential Therapy and Triple Therapy as Second Line Therapy for Refractory Helicobacter Pylori Infection- A Multi-center Randomized Trial
Brief Title: Comparison of the Efficacy of Levofloxacin-based Sequential Therapy and Triple Therapy as Second Line Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: E-DA Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, National Taiwan University Hospital, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201110021MD
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Eradication Rate for Helicobacter
Keywords: H pylori eradication
MeSH Terms: interventions — Lansoprazole; Metronidazole; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- levofloxacin-based sequential therapy (Experimental): levofloxacin-based sequential therapy
  Interventions: Drug: levofloxacin-based sequential therapy
- levofloxacin-based triple therapy (Active Comparator): levofloxacin-based triple therapy for 10 days
  Interventions: Drug: levofloxacin-based triple therapy for 10 days

INTERVENTIONS:
Drug: levofloxacin-based sequential therapy — levofloxacin-based sequential therapy for 10 days〔lansoprazole 30mg and amoxicillin 1g for the first 5 days, followed by lansoprazole 30mg, levofloxacin 250mg, and metronidazole 500mg for another 5 days (all given twice daily)〕
  Other Names: Takepron; Cravit; Flagyl; Amoxicillin
  Arms: levofloxacin-based sequential therapy
Drug: levofloxacin-based triple therapy for 10 days — lansoprazole 30mg and amoxicillin 1g, and levofloxacin 250mg for 10 days (all given twice daily)
  Other Names: Takepron; Cravit; Amoxicillin
  Arms: levofloxacin-based triple therapy

SUMMARY:
To compare the efficacy and tolerability of levofloxacin-based sequential therapy and triple therapy in the second line therapy for those who fail from one eradication therapy

DETAILED DESCRIPTION:
About 600 patients who failed from first line triple therapy or sequential therapy will be eligible in this multicenter randomized comparative trial. Eligible patients will be randomized to receive either (1) levofloxacin-based sequential therapy for 10 days〔lansoprazole 30mg and amoxicillin 1g for the first 5 days, followed by lansoprazole 30mg, levofloxacin 250mg, and metronidazole 500mg for another 5 days (all given twice daily)〕or (2) levofloxacin-based triple therapy for 10 days〔lansoprazole 30mg and amoxicillin 1g, and levofloxacin 250mg for 10 days (all given twice daily)〕. Eradication will be confirmed with 13C-Urea Breath Test 6 weeks after therapy.

ELIGIBILITY:
Inclusion Criteria:

* H. pylori infected patients who failed from first line therapy will be eligible in this study

Exclusion Criteria:

* Patients were excluded from the study if any one of the following criteria was present:
* children and teenagers aged less than 20 years,
* history of gastrectomy,
* gastric malignancy, including adenocarcinoma and lymphoma,
* previous allergic reaction to antibiotics (amoxicillin, metronidazole, levofloxacin) and PPI (lansoprazole),
* contraindication to treatment drugs,
* pregnant or lactating women, or
* severe concurrent disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-12 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Eradication rate in the second line therapy | 6 weeks
  Assessed by UBT

SECONDARY OUTCOMES:
Incidence of adverse effect | 2 weeks
  during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Ming Liou, MD, Principal Investigator — National Taiwan University Hospital
Locations (10):
- Taiwan (10):
  - National Taiwan University Hospital, Hsinchu Branch, Hsinchu
  - E-DA Hospital and I-Shou University, Kaohsiung City
  - Kaohsiung Medical University, Kaohsiung City
  - Health Bureau of Lienchiang County, Lienchiang
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veteran General Hospital, Taipei
  - Mackay Memorial Hospital, Taitung Branch
  - National Taiwan University Hospital , Yunlin, Yunlin

REFERENCES:
- [Background] Liou JM, Chen CC, Chen MJ, Chang CY, Fang YJ, Lee JY, Sheng WH, Wang HP, Wu MS, Lin JT. Empirical modified sequential therapy containing levofloxacin and high-dose esomeprazole in second-line therapy for Helicobacter pylori infection: a multicentre clinical trial. J Antimicrob Chemother. 2011 Aug;66(8):1847-52. doi: 10.1093/jac/dkr217. Epub 2011 May 31. PMID 21632579
- [Derived] Liou JM, Bair MJ, Chen CC, Lee YC, Chen MJ, Chen CC, Tseng CH, Fang YJ, Lee JY, Yang TH, Luo JC, Wu JY, Chang WH, Chang CC, Chen CY, Chen PY, Shun CT, Hsu WF, Hung HW, Lin JT, Chang CY, Wu MS; Taiwan Gastrointestinal Disease and Helicobacter Consortium. Levofloxacin Sequential Therapy vs Levofloxacin Triple Therapy in the Second-Line Treatment of Helicobacter pylori: A Randomized Trial. Am J Gastroenterol. 2016 Mar;111(3):381-7. doi: 10.1038/ajg.2015.439. Epub 2016 Feb 2. PMID 26832653